CLINICAL TRIAL: NCT00884715
Title: Open Label Study to Evaluate the Pharmacokinetics, Efficacy and Safety of Two Doses of an Octreotide Implant in Patients With Carcinoid Syndrome
Brief Title: Pharmacokinetics, Efficacy and Safety of an Octreotide Implant in Patients With Carcinoid Syndrome
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Program was terminated for business reasons
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IP107-002
Record Dates: First submitted 2009-04-20; First posted 2009-04-21 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Carcinoid Syndrome
MeSH Terms: conditions — Serotonin Syndrome | interventions — Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 implant (Experimental): 117 mg Octreotide implant
  Interventions: Drug: Octreotide
- 2 implants (Experimental): 234 mg Octreotide implant
  Interventions: Drug: Octreotide

INTERVENTIONS:
Drug: Octreotide — short acting octreotide

SUMMARY:
Evaluate the pharmacokinetics, safety and efficacy of an octreotide implant for the treatment of the symptoms of carcinoid syndrome.

DETAILED DESCRIPTION:
This study will evaluate a longer acting octreotide formulation. A subcutaneous implant at 2 doses will be evaluated for pharmacodynamics, efficacy and safety for a period of 9 months.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed tumor
* documented evidence of carcinoid syndrome
* life expectancy of at least 6 months
* previous positive octreotide scan
* received stable doses of octreotide injections
* performance status of 0-2 on the ECOG performance scale

Exclusion Criteria:

* poorly differentiated or high grade neuroendocrine tumor
* significant cv, hepatic, renal or other disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-07; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Assess the effects of 1 or 2 implants on carcinoid syndrome symptoms of flushing and diarrhea | 9 months

SECONDARY OUTCOMES:
safety and tolerability of the implants | 9 months

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Iowa City, Iowa
  - Boston, Massachusetts
  - Burlington, Massachusetts

REFERENCES:
- See also: Click here for more information about this study — http://www.endo.com/